CLINICAL TRIAL: NCT01116973
Title: Reliability of Central Venous Pressure Measurements From Peripherally Inserted Central Catheters vs. Centrally Inserted Central Catheters
Brief Title: Reliability of Central Venous Pressure Measurements
Acronym: CVP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in guidelines by the manufacturer.
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1911
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Hemodynamics; Central Venous Pressure
Keywords: CVP monitoring compared with peripheral monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CICC comparison with PICC (Other): All patients will be having CVP reading taken from the CICC
  Interventions: Other: PICC
- PICC group (Other): The transition to the PICC, a 5.0-French, 18-gauge double lumen PICC (BARD, Power PICC Solo Catheter with Tip Location Stylet; Salt Lake City, UT) will be inserted
  Interventions: Other: PICC

INTERVENTIONS:
Other: PICC — Peripheral inserted catheter placement to take the reading
  Other Names: 18-gauge double lumen PICC

SUMMARY:
The purpose of this study is to compare CVP measurements from CICCs and PICCs. The investigators will also evaluate whether or not the duration of CICC placement affects the differences in CVP measurements between the CICCs and PICCs. The investigators hypothesize that the differences between the CVP measurements of the CICCs and PICCs will be clinically insignificant.

DETAILED DESCRIPTION:
Centrally inserted central catheters (CICC) are commonly used in the intensive care unit (ICU) for delivery of fluids, medications, and nutrition. They are also used to measure central venous pressure (CVP) which provides critical information about blood volume status and cardiac function of a patient. Currently, CICCs are the gold standard for measuring CVP, but they have a number of associated risks including pneumothorax, major hemorrhage, neck hematoma, and carotid puncture. An alternative to a CICC is a peripherally inserted central catheter (PICC). A PICC can be placed with lower risks than a CICC, has a lower rate of bloodstream infections, and provides longer-term IV access at a lower cost. PICCs can be used to deliver fluids, medications, and nutrition. However, there is minimal evidence that a PICC can measure CVP as effectively as a CICC. Therefore, a CICC is preferred when a patient requires CVP monitoring in our ICU. Our aim is to compare CVP measurements from CICCs and PICCs. We will also evaluate whether or not the duration of CICC placement affects the differences in CVP measurements between the CICCs and PICCs. We hypothesize that the differences between the CVP measurements of the CICCs and PICCs will be clinically insignificant.

The goal of this study is to determine if the central venous pressure (CVP) measurements obtained from a peripherally inserted central catheter (PICC) consistently correlate with the CVP measurements obtained from a centrally inserted central catheter (CICC). If the difference between the CVP measurements from the CICC and PICC are found to be clinically insignificant, then it may be practical to place PICCs in favor of CICCs thereby avoiding some of the potential complications associated with CICC placement. We also aim to evaluate whether or not the duration of CICC placement affects the differences in CVP measurements between the CICCs and PICCs. We hypothesize that the differences between the CVP measurements of the CICCs and PICCs will be clinically insignificant.

ELIGIBILITY:
Inclusion Criteria:

* Subject's ability to lay in a supine position with their hands at their sides during CVP measurements
* A consent form signed by the patient or patient's representative
* Subjects that are age 18-90
* Subjects that have an indwelling CICC and are transitioning to a PICC for long-term IV access
* CICC placed in the internal jugular vein or subclavian vein position

Exclusion Criteria:

* Inability to obtain consent
* Subjects under 18 years of age
* Non-English speaking subjects
* Subjects that are unable to lay flat due to pulmonary complications, increased intracranial pressure (ICP), or unstable spinal cord injuries
* Subjects with known cardiac abnormalities (atrial septal defects or ventricular septal defects, severe tricuspid valve disease, severe pulmonary hypertension, Ejection fraction < 15%)
* Prisoners
* Subjects with known upper extremity deep vein thromboses (subclavian or distal)
* Subjects with non-functional CICC or PICC distal ports
* Subjects with femoral CICCs
* Pregnant women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-09-02 (Actual); Primary Completion 2016-08-27 (Actual); Study Completion 2016-08-27 (Actual)

PRIMARY OUTCOMES:
Central venous pressure comparison with peripheral venous pressure | 1 year
  We will compare the realiablity of reading collected via central venous pressure reading and compare it with peripheral venous pressure reading.

SECONDARY OUTCOMES:
CICC reading comparison with PICC | 1 year
  This might also reduce the complications associated with CICC procedures

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Roberts, MD, Principal Investigator — University of Oklahoma
Locations (2):
- United States (2):
  - Univeristy of Oklahoma Health Sciences Center Dept. Anesthesiology, Oklahoma City, Oklahoma
  - Univeristy of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No